CLINICAL TRIAL: NCT06570928
Title: Use of a Product Containing the Cannabinoids CBD and THC as a Treatment Strategy for Alzheimer's Disease - Clinical Trial Alzheimer's Disease and Cannabis (DAZACANN)
Brief Title: Use of a Cannabinoids as a Treatment Strategy for Alzheimer's Disease
Acronym: DAZACANN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Latin American Integration (Other)
Responsible Party: Principal Investigator, FRANCISNEY PINTO DO NASCIMENTO, Professor and Coordinator of the Laboratory of Medicinal Cannabis and Psychedelic Science, Federal University of Latin American Integration
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAZACANN
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Cannabinoids; Cannabidiol; Tetrahydrocannabinol (THC); Nervous System Diseases
MeSH Terms: conditions — Alzheimer Disease; Nervous System Diseases | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: 72 patients will be randomized into 2 groups. One group will receive a product containing CBD/THC and the other group will receive a placebo, a compound with the same characteristics, without an active ingredient.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and caregivers will not know what they are using. The investigators evaluating it won't know either. Only a team member who is not part of the investigative team will know.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo arm (Placebo Comparator): Patients will receive a liquid solution only with vehicle and no cannabinoid.
  Interventions: Other: Placebo
- Experimental arm (Experimental): Patients will receive the dose of 0,2 ml of a compound contain CBD:THC (50 mg:5 mg).
  Interventions: Other: Cannabis

INTERVENTIONS:
Other: Cannabis — 0,2 ml of CBD:THC (50 mg:5 mg)
  Other Names: CBD:THC (50 mg:5 mg)
  Arms: Experimental arm
Other: Placebo — Product vehicle, medium chain triglycerides (MCT)
  Arms: Placebo arm

SUMMARY:
Brief Summary:

The objective of the study is to evaluate the effect of cannabinoids on Alzheimer's Disease. This is a double-blind, randomized, placebo-controlled clinical trial. The study aims to recruit patients of both sexes diagnosed with Alzheimer's Disease who are in the mild and moderate stages for treatment with cannabinoids.

The specific objectives of the study are:

Primary Outcome

* To evaluate the effect of Cannabis sativa at low doses according to the Mini-Mental State Examination (MMSE) scale - Memory and Cognition test - in patients with Alzheimer's Disease.

Secondary Outcomes

* To evaluate the effect of Cannabis sativa at low doses according to the Cornell scale - Depression in dementia test.
* To evaluate the effect of Cannabis sativa at low doses according to the GDS scale - Depression in elderly people test.
* To evaluate the effect of Cannabis sativa at low doses according to the QoL scale - Quality of Life test.
* To evaluate the effect of Cannabis sativa at low doses according to the Epworth scale - Drowsiness test.
* To evaluate the adverse effects of Cannabis sativa at low doses given daily for 26 weeks in patients with Alzheimer's Disease.

Participants will use a compound containing CBD/THC 50/5 mg/mL, administered as 0.2 mL once a day. The placebo group will use a compound identical to the treatment but containing only vehicle. To address the questions above, the treated group will be compared with the placebo group over a period of 6 months. Participants will be assessed every 2 months. Additionally, blood and cerebrospinal fluid tests will be conducted to measure specific proteins related to Alzheimer's Disease and inflammatory markers.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is closely linked to the accumulation of neurotoxins derived from Aβ and tau, leading to cognitive impairment. This project posits that an imbalance in the endocannabinoid system occurs in an AD-dependent manner. Reported connections between dementia, inflammation, Aβ, and alterations in the cannabinoid system in experimental models of AD support this hypothesis. Cannabinoids may restore baseline brain function while avoiding major side effects. Despite extensive research into new AD therapies, no significant improvement has been achieved recently, and there is little consensus on how scientists will innovate to develop a new treatment. Cannabinoid-based therapy has emerged as crucial for the treatment of many diseases considered incurable. The expected results of this project will provide important insights into the ability of cannabinoids to counteract neurochemical imbalance during AD progression, thereby improving memory performance and affecting inflammation as well as Aβ and tau levels.

The key point is to provide evidence that cannabinoids can serve as an efficient treatment for AD while avoiding major side effects. The aim of this project is to determine the effect of cannabinoids in AD patients, evaluating memory and cognition. It is expected that the results will establish that cannabinoids are critical for restoring the baseline function of the endocannabinoid system in AD brains and their beneficial effects. This project may be instrumental in validating new therapeutic approaches for AD.

To evaluate the pharmacological activity of low doses of CBD, a double-blind, randomized, placebo-controlled clinical trial will be conducted for a duration of 6 months. A baseline assessment will be performed, and patients will be evaluated every 60 days for a period of 6 months, totaling 4 evaluation sessions. For this purpose, the following questionnaires will be applied: Mini-Mental State Examination (MMSE), Neuropsychiatric Inventory (NPI), Geriatric Depression Scale (GDS), Alzheimer's Disease Quality of Life version patient, version caregiver and caregiver-patient version, Cornell Depression in Dementia Scale, and Epworth Sleepiness Scale. All questionnaires are references in their assessment domains and are validated for Portuguese/Brazil. In addition to the evaluation scales, biological material will be collected with blood and cerebrospinal fluid samples at baseline and at the end (after 6 months). The following analytes will be measured in the CSF: BDNF, beta-amyloid, Tau protein, TNFα, IL-6, IL-1β, and IL-10. During the research and data collection, patients' conventional treatments will not be altered.

Statistical Analysis Plan SPSS software, version 29.0 will be used for the analyses. For quantitative data, the Shapiro-Wilk distribution test will be performed. Potential associations between qualitative variables will be analyzed using the Chi-Square test with adjusted residual analysis (χ²). The means (±SD) will be analyzed using the Student's t test for independent samples. Medians [IQR] will be calculated using the Mann-Whitney U test. Paired quantitative data will be compared individually by group across the analyzed time points using Friedman's ANOVA test.

A generalized estimating equations (GEE) model, linear or with log-gamma link, and Bonferroni correction will be used to simultaneously evaluate quantitative parameters over time and between groups. For these descriptive analyses, data will be presented as means ± standard errors (±SEM). Pearson or Spearman correlations can be performed between variables of interest. For all analyses, the significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Be over 60 years old;
* Have been diagnosed with AD at least 1 year ago;
* Present mild to moderate symptoms of AD.

Exclusion Criteria:

* Have a diagnosis of other dementias or factors correlated;
* Present psychosis or first-degree relatives with a history from psychosis, schizophrenia, epilepsy;
* Individuals with a history of psychoactive substance abuse will be included in the study;
* Present severe symptoms of AD.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Exam (MMSE) | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  scores range from 0 to 30, with higher scores indicating cognitive improvement.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory-Questionnaire (NPI-Q) | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  Assesses neuropsychiatric symptoms in patients with dementia. Evaluates 12 symptoms in the following domains: delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor behaviors, nocturnal behavioral disorders, and appetite disorders. The score ranges from 0 to 144.
Geriatric Depression Scale (GDS) | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  Assesses depressive symptoms in the elderly. The investigators will use the short version, which has a score from 0 to 15. The higher the score, the greater the depressive symptoms.
Quality of Life in Alzheimer's Disease scale (QoL-AD) | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  The scale has 3 versions, one of which is applied to the patient, another to the caregiver to answer about the patient's life, and one for the caregiver to answer about their own life. The score may vary, the one the investigators will use is the sum of the questionnaires about the patient, caregiver version and patient version, with the patient version having a weight of 2. Its score varies from 13, indicating the worst possible quality of life, up to 52, and the higher the score, the higher the quality of life.
Cornell Scale for Depression in Dementia (CSDD) | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  Assess symptoms of depression in patients with dementia. Has 19 questions applied to caregiver and patient. The maximum score is 38 points, with scores higher than 10 indicating probable major depression and greater than 18 as major depression.
Epworth Sleepiness Scale (ESS ) | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  Evaluates 8 items with scores ranging from 0 to 24, in which scores higher than 10 indicate sleep disturbances.
Specific markers of Alzheimer's disease: Beta-amyloid 40, beta-amyloid 42, tau protein (fraction 181), and phosphorylated tau protein | Collections will be made at the initial time, before the start of treatment and at the end time, after 180 days.
  The following proteins will be quantified in the cerebrospinal fluid: beta-amyloid 40, beta-amyloid 42, tau protein (fraction 181), and phosphorylated tau protein.
BDNF (Brain Derived Neurotrophic Factor) | Collections will be made at the initial time, before the start of treatment and at the end time, after 180 days.
  It will be measured in serum or plasma
Inflammatory markers: TNFα (Tumor Necrosis Factor alpha), IL-6 (Interleukin-6), IL-1β (Interleukin-1 beta), and IL-10 (Interleukin-10) | Collections will be made at the initial time, before the start of treatment and at the end time, after 180 days.
  It will be measured in serum or plasma

OTHER OUTCOMES:
Safety Endpoints - UKU Side Effect Rating Scale | The participants will be evaluated before starting treatment, and then every 60 days until 180 days are complete, resulting in 4 evaluations.
  Will be conducted on patients and caregivers during all planned visits to ascertain the frequency and severity of adverse events. There will be neurological and physical examinations as well as laboratory testing.

CONTACTS AND LOCATIONS:
Overall Officials: Taynara Silva, 1, Principal Investigator — Universidade Federal de Santa Catarina
Locations (1):
- Federal University of Latin American Integration, Foz do Iguaçu, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No